CLINICAL TRIAL: NCT03745885
Title: A Randomized, Double-blind, Placebo-controlled Study the Efficacy and Safety of Supaglutide in Chinese Healthy Subjects
Brief Title: A Study of the Efficacy and Safety of Supaglutide in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Yinnuo Pharmaceutical Technology Co., Ltd. (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YN011A
Record Dates: First submitted 2018-11-16; First posted 2018-11-19 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 0.15mg Supaglutide or placebo (Experimental): 0.15 milligrams (mg) Supaglutide injection or placebo administered once subcutaneously（SC） to healthy participants
  Interventions: Drug: Supaglutide injection; Drug: Placebo
- 0.375mg Supaglutide or placebo (Experimental): 0.375 milligrams (mg) Supaglutide injection or placebo administered once subcutaneously（SC） to healthy participants
  Interventions: Drug: Supaglutide injection; Drug: Placebo
- 0.75mg Supaglutide or placebo (Experimental): 0.75 milligrams (mg) Supaglutide injection or placebo administered once subcutaneously（SC） to healthy participants
  Interventions: Drug: Supaglutide injection; Drug: Placebo
- 1.5mg Supaglutide or placebo (Experimental): 1.5 milligrams (mg) Supaglutide injection or placebo administered once subcutaneously（SC） to healthy participants
  Interventions: Drug: Supaglutide injection; Drug: Placebo
- 3.0mg Supaglutide or placebo (Experimental): 3.0 milligrams (mg) Supaglutide injection or placebo administered once subcutaneously（SC） to healthy participants
  Interventions: Drug: Supaglutide injection; Drug: Placebo

INTERVENTIONS:
Drug: Supaglutide injection — Administered SC in the Supaglutide arms.
  Other Names: Diabegone
Drug: Placebo — Administered SC in the placebo arms and to maintain the blind in the Supaglutide injection arms.

SUMMARY:
This study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of the investigational drug Supaglutide proposed dosing once (or twice) weekly in Chinese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects between 18 and 45 years old（inclusive）.
2. Body mass index（BMI）is between 18 and 28 kg/m2 (inclusive). The weight of male subjects should not be less than 50 kg, and female subjects should not be less than 45 kg.
3. The female participant with reproductive potential, will be required a negative pregnancy test before trial, maintaining non-pregnancy during the whole study period and contraception 3 months after formal injection.
4. Participants must sign the informed consent.

Exclusion Criteria:

1. Have a history of allergic reaction or hypersensitivity to the study drugs, or who develop allergic reaction.
2. Have an evidence of Fasting blood-glucose greater than (>) 6.0 mmol/L or less than (<) 3.9 mmol/L, or hemoglobin A1c (HbA1c) greater than or equal to (>=) 6.5 percent (%);
3. Have evidence of Sitting Blood ( take a break for five minutes) , systolic pressure exceeds the range of 90 to 140 mmHg, or diastolic pressure exceeds the range of 50 to 90 mmHg, or Heart Rate exceeds the range of 50 bpm to100 bpm (including critical value)
4. Have an evidence of ECG abnormalities including QTc >450 msec or QRS complex >120 msec. If QT Corrected >450 msec; or QRS >120msec, subject should Repeat the ECG measurements twice and use the average of the QTc or QRS values measured to determine whether the subjects are eligible.
5. Have an evidence of physical examination, vital sign, laboratory examination or electrocardiographic examination that investigator think can affect this trial;
6. Have an individual or a family history of thyroid C-cell tumors/ carcinoma or with a history of thyroid dysfunction, thyroid hormone abnormalities or thyroid-related hormones exceeded the normal range;
7. Have a history of significant illness or medical disorders, including acute or chronic pancreatitis, cardiovascular disease, renal disorder, hematological disease，hepatic or gastrointestinal disease, neurological or psychiatric disease, metabolic disorder, or other diseases that may affect the absorption, distribution, metabolism or excretion of drugs, such as active gastrointestinal ulcers or bleeding, gastrointestinal surgery(except appendectomy).
8. Have a history of major surgery within 4 weeks or major minor surgery during the whole study period;
9. Have a history of smoking or the use of nicotine products or electronic cigarettes, abusing alcohol or abusing drug within 3 months;
10. Have a presence of prescription or non-prescription drugs, including Chinese Traditional and Herbal Drugs within 2 weeks; Previous use of glucagon-like peptide-1 analogue or another intestinal insulin, or any unknown cause of infections.
11. Have a presence of any food or drink containing caffeine or xanthine within 48 hours before administration.
12. Have a history of a New Chemical Entity clinical study within the previous 3 months.
13. Have a presence of pregnancy or lactation.
14. Have a presence of positive hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV), or human immunodeficiency virus (HIV) antibody, or treponema pallidum antibody.
15. Have a history of blood donation or loss more than 400 ml (including in the frame of a clinical study) within 3 months before administration;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic：Cmax of Supaglutide | baseline and up to 29 days after formal dose
  Maximum Concentration(Cmax) of Supaglutide
Pharmacokinetic: Tmax of Supaglutide | baseline and up to 29 days after formal dose
  Time to maximum plasma concentration (Tmax)
Pharmacokinetic: AUC0-t of Supaglutide | baseline and up to 29 days after formal dose
  Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC0-t)
Pharmacokinetic: t½ of Supaglutide | baseline and up to 29 days after formal dose
  Terminal elimination half-life in plasma (t½)

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lou YR, Xu YL, Xiong Y, Deng C, Wang Q. Population Pharmacokinetics of Efsubaglutide Alfa in Healthy Subjects and Subjects with Type 2 Diabetes. Clin Pharmacokinet. 2025 Apr;64(4):533-552. doi: 10.1007/s40262-025-01475-7. Epub 2025 Feb 17. PMID 39961992